CLINICAL TRIAL: NCT02064036
Title: Whole-Pelvic Radiotherapy With a Stereotactic Body Radiotherapy Boost and Long-Term Androgen Deprivation for Unfavorable-Intermediate and High Risk Localized Adenocarcinoma of the Prostate.
Brief Title: Stereotactic Boost and Long-Term Androgen Deprivation for Adenocarcinoma of the Prostate
Acronym: CCRO025
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of California, Davis (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 421870; CCRO025 (Other: UC Davis)
Record Dates: First submitted 2014-01-22; First posted 2014-02-17 (Estimated); Last update posted 2022-10-18 (Actual); Status verified 2022-10

CONDITIONS: Adenocarcinoma of the Prostate
Keywords: Prostate Cancer; Radiotherapy; Androgen Deprivation
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Radiotherapy, Intensity-Modulated; Radiotherapy; X-Ray Therapy; Radiation; bicalutamide; Leuprolide; Goserelin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Single (Experimental): Neoadjuvant Androgen Blockade (Casodex) Followed by: Intensity Modulated Radiotherapy (IMRT)2 with Concurrent Androgen Blockade (Casodex and Leuprolide) to Whole Pelvis, Prostate, and Seminal VesiclesFollowed by: Stereotactic Radiosurgical Boost3 to the Prostate with Implanted Electromagnetic Transponder Beacon Intrafraction Guidance Followed by: Adjuvant Androgen Blockade (Casodex)
  Interventions: Radiation: Stereotactic Radiosurgical Boost; Drug: Casodex; Drug: Leuprolide

INTERVENTIONS:
Radiation: Stereotactic Radiosurgical Boost — Intensity Modulated Radiotherapy (IMRT)2 with Concurrent Androgen Blockade to Whole Pelvis, Prostate, and Seminal Vesicles Followed by: Stereotactic Radiosurgical Boost3 to the Prostate with Implanted Electromagnetic Transponder Beacon Intrafraction Guidance
  Other Names: Intensity Modulated Radiotherapy (IMRT); Radiotherapy,; X-ray therapy; Irradiation
Drug: Casodex — Neoadjuvant Androgen Blockade before radiation therapy and Adjuvant Androgen Blockade after radiation therapy
  Other Names: Bicalutamide
Drug: Leuprolide — Neoadjuvant Androgen Blockade before radiation therapy and Adjuvant Androgen Blockade after radiation therapy
  Other Names: Goserelin

SUMMARY:
We hypothesize that Stereotactic Body Radiotherapy Boost (SBRT) as a boost to the prostate following whole pelvic intensity modulated radiotherapy (IMRT) can be delivered effectively and safely in a population of men with unfavorable intermediate and high risk localized prostate cancer.

Our primary objective is to assess the feasibility and safety of a treatment strategy incorporating whole pelvic IMRT followed by an SBRT boost to the prostate with neoadjuvant, concurrent, and adjuvant androgen deprivation for a total of 28 months for men with unfavorable intermediate or high risk localized prostate cancer.

DETAILED DESCRIPTION:
The primary objective of this study is to assess the feasibility and safety of a treatment strategy incorporating whole pelvic IMRT followed by an SBRT boost to the prostate with neoadjuvant, concurrent, and adjuvant androgen deprivation for a total of 28 months for men with unfavorable intermediate or high risk localized prostate cancer.

The secondary objective is to assess biochemical control at 24 months following the experimental treatment strategy by the "Phoenix definition". Patients not meeting these prostate-specific antigen (PSA) criteria (Phoenix Definition) for failure who undergo salvage therapies (such as androgen deprivation therapy (ADT), radical prostatectomy or brachytherapy, or Cryosurgery) should also be declared as failures at the time a positive biopsy is obtained or salvage therapy is administered, whichever comes first.

Another secondary objective is to assess toxicity of the experimental treatment approach as scored by the Common Terminology Criteria for Adverse Events The third secondary objective is to assess prostate organ motion during hypofractionated radiotherapy. To assess motion of the prostate during the protracted delivery of hypofractionated radiotherapy as assessed by implanted electromagnetic transponder beacons.

ELIGIBILITY:
Inclusion Criteria:

1. Pathologically (histologically or cytologically) proven diagnosis of prostatic adenocarcinoma within 180 days of registration at moderate to high risk for recurrence
2. History/physical examination (to include at a minimum digital rectal examination of the prostate and examination of the skeletal system and abdomen) within 90 days prior to registration.
3. Clinically negative lymph nodes as established by imaging (pelvic ± abdominal CT or MRI), (but not by nodal sampling, or dissection) within 90 days prior to registration.
4. Patients with lymph nodes equivocal or questionable by imaging are eligible if the nodes are ≤ 2.0 cm.
5. No evidence of bone metastases (M0) on bone scan within 90 days prior to registration.
6. Equivocal bone scan findings are allowed if plain films (or CT or MRI) are negative for metastasis.
7. Baseline serum PSA value performed with an FDA-approved assay (e.g., Abbott, Hybritech) within 12 weeks (90 days) prior to registration.
8. Study entry PSA should not be obtained during the following time frames: (1) 10-day period following prostate biopsy; (2) following initiation of hormonal therapy; (3) within 30 days after discontinuation of finasteride; (4) within 90 days after discontinuation of dutasteride.
9. Zubrod Performance Status 0-2
10. Complete blood count (CBC)/differential obtained within 2 weeks (14 days) prior to registration on study, with adequate bone marrow function
11. Patient must be able to provide study specific informed consent prior to study entry.

Exclusion Criteria:

1. Prior invasive (except non-melanoma skin cancer) malignancy unless disease-free for a minimum of 2 years.
2. Previous radical surgery (prostatectomy) or cryosurgery for prostate cancer
3. Previous pelvic irradiation, prostate brachytherapy, or bilateral orchiectomy
4. Previous hormonal therapy
5. Prior pharmacologic androgen ablation for prostate cancer is allowed only if the onset of androgen ablation is ≤ 60 days prior to the date of registration.
6. Use of finasteride within 30 days prior to registration
7. Use of dutasteride or dutasteride/tamsulosin (Jalyn) within 90 days prior to registration
8. Previous or concurrent cytotoxic chemotherapy for prostate cancer; note that prior chemotherapy for a different cancer is allowable. See Section 3.2.1.
9. Prior radiotherapy, including brachytherapy, to the region of the study cancer that would result in overlap of radiation therapy fields
10. Severe, active co-morbidity including heart issues, infection and liver problems
11. Patients who are sexually active and not willing/able to use medically acceptable forms of contraception
12. Prior allergic reaction to the hormones involved in this protocol
13. Patients status-post a negative lymph node dissection are not eligible

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2013-06-06 (Actual); Primary Completion 2020-12-03 (Actual); Study Completion 2021-10-29 (Actual)

PRIMARY OUTCOMES:
Tumor Assessment | 24 months
  Tumors will be assessed using the American Joint Committee on Cancer (AJCC) Staging System, 7th Edition. This system consists of the following subscales: the extent of the primary tumor (T category), whether the cancer has spread to nearby lymph nodes (N category), the absence or presence of distant metastasis (M category), the PSA level at the time of diagnosis, and the Gleason score, based on the prostate biopsy (or surgery).

SECONDARY OUTCOMES:
Zubrod Performance Scale | Weekly during radiation treatment; every three months during hormone therapy; every six months for 3 yrs after hormone therapy
  This is a scale used to evaluate the patient's performance status is an attempt to quantify cancer patients' general well-being and activities of daily life.

CONTACTS AND LOCATIONS:
Overall Officials: Richard Valicenti, MD, Principal Investigator — University of California, Davis
Locations (1):
- UC Davis Sacramento Cancer Center Dept of Radiation Oncology, Sacramento, California, United States

IPD SHARING:
Plan to Share IPD: No